CLINICAL TRIAL: NCT01988688
Title: Pilot Study of Deep Brain Stimulation (DBS)in Area LC for Chronic Tinnitus
Brief Title: Pilot Study of Deep Brain Stimulation (DBS) in Area LC for Chronic Tinnitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paul Larson (Other)
Responsible Party: Sponsor-Investigator, Paul Larson, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBS Tinnitus
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Tinnitus
Keywords: deep brain stimulation
MeSH Terms: conditions — Tinnitus | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bilateral DBS placement in area LC (Experimental): Bilateral DBS placement in area LC. Devices include Medtronic Activa DBS model 3387 and 3389; Medtronic DBS extension; Medtronic Activa PC or Activa RC neurostimulator; Medtronic Patient Programmer; Medtronic Test Stimulator; Medtronic N/Vision Clinician Programmer
  Interventions: Device: Deep Brain Stimulation (DBS)

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) — Deep Brain Stimulation (DBS) bilaterally in area LC.

SUMMARY:
This study will test the safety and effectiveness of deep brain stimulation (DBS) for patients with a big or very big problem with tinnitus (a sensation of noise in the head).

DETAILED DESCRIPTION:
This is a single institution, open-label, phase I clinical trial to estimate the treatment effect size and to assess preliminary safety and tolerability of DBS in the caudate nucleus (area LC) in adults with a big or very big problem (tinnitus functional index TFI>50) with chronic tinnitus. Up to 10 subjects will be implanted. The DBS stimulation parameters are patient-specific and will be allowed to vary over the course of the treatment periods, calibrated by the TFI. During Period I, stimulation will be continuous. During Period II, there will be three stimulation OFF/ON epochs, where the stimulation will be turned OFF and then turned back ON when the tinnitus loudness returns to a certain level (based on a change in the TFI score). During Period III, stimulation will be "on demand," i.e. controlled by the subject and determined by subject preference. An important goal is to determine whether tinnitus can be controlled through optimization of stimulation parameters.

ELIGIBILITY:
Inclusion Criteria:

Men and women between the ages of 22 and 75 years. Subjective, unilateral or bilateral, non-pulsatile tinnitus of 1 year's duration or greater.

Tinnitus Functional Index (TFI) score greater than 50. Tinnitus unresponsive acoustical and behavioral therapies. Prospective subjects must have received at least one acoustical (masker, hearing aid, Neuromonics®) or behavioral therapy (cognitive behavioral, directive counseling, tinnitus retraining therapy) to be eligible for study enrollment, but partial response to conventional therapy does not exclude a prospective subject if the individual meets the TFI > 50 study participation threshold.

Montreal Cognitive Assessment (MoCA) ≥ 26. Subjects of child-bearing potential using an appropriate form of birth control acceptable to the research team and with a negative urine pregnancy test or has undergone sterilization procedure.

Capacity to give informed consent. English-speaking.

Exclusion Criteria:

Patients experiencing tinnitus related to untreated retrocochlear lesion, or other known anatomic/structural lesions of the ear or temporal bone.

Patients with hyperacusis or misophonia (hypersensitivity to loud noises). Hearing loss of moderately severe or greater severity in either ear. History of seizure disorder or currently under treatment for seizure disorder. Patients with cardiac pacemakers, intracardiac lines, implanted medication pumps, implanted electrodes in the brain, other intracranial metal objects with the exception of dental fillings, or any other contraindication for obtaining a MRI scan.

Patients with an acute or chronic unstable medical condition which, in the opinion of the PI, would require stabilization prior to or preclude DBS surgery.

Patients with any active ear disease that, in the opinion of the PI, needs to be further evaluated.

Patients with psychiatric symptoms that, in the opinion of the study team, are not adequately treated or would interfere with study activities.

Any psychiatric co-morbidity that may complicate the interpretation of study results.

Pregnancy. Currently breast-feeding. Patients with tinnitus related to Workman's Compensation claim or litigation-related event.

Patients taking any medication(s), in the opinion of the PI, that is (are) deemed to be etiologically related to the development of tinnitus.

Preoperative neurophychological evaluation that indicates either of the following:

Dementia - Using DSM-IV criteria of memory impairment and at least one of the following: aphasia, apraxia, agnosia or disturbances in executive functioning. The cognitive impairments must be severe enough to cause impairment in social and occupational functioning and must represent a decline from a previously higher level of functioning. The diagnosis of dementia will not be made if the cognitive deficits occur exclusively during the course of a delirium.

Cognitive impairment (z < -1.5) in multiple domains without dementia (i.e. patient is functionally intact), but in the opinion of the study team would not or could not comply with study requirements.

Beck Depression Inventory-II (BDI-II) > 29, indicating severe depression. Patients with a history of claustrophobia that would interfere with MRI or surgery.

Active alcohol and/or drug dependence or history of alcohol and/or ETOH dependence within the last year.

Any medical condition that, in the opinion of the investigators, confounds study results or places the subject at greater risk.

Unable to provide informed consent.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Tinnitus Functional Index (TFI) score change | Up to 18 months
  Between Baseline and Period I, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Paul Larson, MD, Principal Investigator — San Francisco VA Medical Center; Steven Cheung, MD, Principal Investigator — San Francisco VA Medical Center
Locations (1):
- San Francisco Veterans' Administration Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Cheung SW, Racine CA, Henderson-Sabes J, Demopoulos C, Molinaro AM, Heath S, Nagarajan SS, Bourne AL, Rietcheck JE, Wang SS, Larson PS. Phase I trial of caudate deep brain stimulation for treatment-resistant tinnitus. J Neurosurg. 2019 Sep 24;133(4):992-1001. doi: 10.3171/2019.4.JNS19347. Print 2020 Oct 1. PMID 31553940
- [Derived] Perez PL, Wang SS, Heath S, Henderson-Sabes J, Mizuiri D, Hinkley LB, Nagarajan SS, Larson PS, Cheung SW. Human caudate nucleus subdivisions in tinnitus modulation. J Neurosurg. 2019 Feb 8;132(3):705-711. doi: 10.3171/2018.10.JNS181659. Print 2020 Mar 1. PMID 30738400